CLINICAL TRIAL: NCT03072251
Title: Participation of Breast Milk Feeding Mothers in Research
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Leanne Redman, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 2017-006
Record Dates: First submitted 2017-02-24; First posted 2017-03-07 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Breastfeeding; Energy Intake; eHealth
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anyone: Any individual may complete this survey

SUMMARY:
To assess concerns and barriers for measuring milk intake of breast fed infants using the remote food photography method and SmartIntake smartphone application. These data will 1) provide support for further development of the Infant RFPM and 2) provide important preliminary data in a National Institutes of Health grant application being developed and assess the prevalence of exclusive breastfeeding and complementary breastfeeding in the study population.

DETAILED DESCRIPTION:
Study participation will be the completion of an anonymous, online survey powered by HIPAA compliant REDCap database. The survey will be made available to potential participants through the internet. The survey will take approximately five minutes to complete. The expected duration of recruitment and completion of the study is six months.

ELIGIBILITY:
Inclusion Criteria:

* Any individual may take the survey.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from the community via print, electronic, and social media. Any individual may take the survey.
Sampling Method: Non-Probability Sample
Enrollment: 570 (Actual)
Dates: Start 2017-02-05 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Receptivity for measuring milk intake for 5-7 days using a smartphone app | 1 day
  Outcome measured by questionnaire

SECONDARY OUTCOMES:
Receptivity for expressing human breast milk to assess milk intake for 5-7 days | 1 day
  Outcome measured by questionnaire

OTHER OUTCOMES:
Prevalence of breastfeeding in the survey population (exclusive, in combination with infant formula, in combination with other foods) | 1 day
  Outcome measured by questionnaire
Method of feeding (breast, expressed human milk in an infant feeding bottle, combination of feeding methods) | 1 day
  Outcome measured by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Redman, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No